CLINICAL TRIAL: NCT02529592
Title: Endotoxin-induced Inflammatory and Behavioral Responses and Predictors of Individual Differences: A Randomized, Double-blind Placebo Controlled Study on Healthy Human Volunteers
Brief Title: Endotoxin-induced Inflammatory and Behavioral Responses and Predictors of Individual Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Mats Lekander, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: LPS 2.0 - 2014/1946-31
Record Dates: First submitted 2015-04-29; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Sickness Behavior
Keywords: Sickness behavior; Cytokines; Psychoneuroimmunology
MeSH Terms: conditions — Illness Behavior | interventions — Endotoxins; Lipopolysaccharides; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotoxin (Experimental): Endotoxin at 2ng/kg of body weight administered intravenously
  Interventions: Biological: Endotoxin
- Placebo (Placebo Comparator): Placebo administered intravenously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Endotoxin
  Other Names: LPS; lipopolysaccharide
  Arms: Endotoxin
Biological: Placebo
  Other Names: NaCl 0.9%; saline
  Arms: Placebo

SUMMARY:
The objective of the present study is to specifically assess the effect of lipopolysaccharide (LPS) administration on the development of behavioral symptoms and the underlying contribution of inflammatory processes. In particular, the investigators will assess the development of subjective and objective behavioral symptoms. In addition, the investigators will determine whether some psychological trait or state can predict and/or modulate the LPS-induced inflammatory and behavioral responses.

Twenty-five healthy subjects will be included. A placebo-controlled, double-blinded and cross-over design will be used. Subjects will receive an intravenous injection of endotoxin at 2 nanogram/kilogram (ng/kg) of body weight and an intravenous injection of sodium chloride as placebo of endotoxin injection at two different occasions.

Prior to inclusion and randomization, subjects will come at the hospital and will receive a medical examination. Psychological variables that could affect the behavioral (or immune) response to LPS will be assessed at that time, using several self-assessment questionnaires.

On the trial days, injection of endotoxin or sodium chloride will be performed and blood samples will be taken just before the endotoxin or sodium chloride injection and 1, 1.5, 2, 3, 4, 5, 6 and 7.5 hours after the injection. Blood samples will be used to measure several inflammatory and immune markers. Urine samples will be taken before the endotoxin or sodium chloride injection and as late as possible after the injection. Subjects will wear T-shirt all day. Urine and T-shirt samples will be used for behavioral assessment and analysis of body odor compound.

Self-assessment questionnaires assessing behavioral and psychological variables will be completed by participants just before the endotoxin or sodium chloride injection, three hours and 7.5 hours after the injection. A short questionnaire assessing sickness behavior (SicknessQ) will be repeatedly completed by participants from just before to 7.5 hours after the endotoxin or sodium chloride injection.

Several behavioral tests will be used, including a motivation task, a test assessing behavioral response to negative and sickness stimuli. Analysis of gait and motion, as well as of social interactions, will be performed. Photographs will be taken for the further rating of the faces.

DETAILED DESCRIPTION:
Study design

Twenty-five subjects will be included in the present study, which will follow a prospective, placebo-controlled and cross-over design. Participants will be blinded, as well as research personnel in charge of the participants and the laboratory.

Subjects will be randomly assigned in the cross-over design with two trials, with about four weeks wash-out between LPS stimulations:

1. Trial 1: endotoxin. Subjects will receive an intravenous injection of endotoxin at 2 ng/kg of body weight.
2. Trial 2: placebo. Subjects will receive an intravenous injection of sodium chloride as placebo of endotoxin injection.

Ten other healthy volunteers will be recruited in a pilot study prior the beginning of the main study, in order to test the behavioral tasks that will be used. These subjects will be recruited among the university staff or among university students. They will perform four specific behavioral tasks and will complete the questionnaires assessing psychological and behavioral variables in order to associate outcomes from the behavioral tasks to psychological and subjective behavioral assessments. No biological samples (blood, urine or tee-shirt samples) will be taken in subjects recruited in the pilot study.

Treatment

The LPS is provided by LGC Promochem AB, Albanoliden 5, 4tr, 506 30 Borås, Sweden. The USP (United States Pharmacopeial Convention) Endotoxin (Cat. No. 1235503) does come as a lyophilized (freeze-dried) powder and each vial contains 10,000 USP Endotoxin Units. Each vial contains very approximately 1 microgram of Endotoxin and is mixed with 5 milliliter (mL) of sterile water.

Study procedure

The study will be conducted at Department of Clinical Sciences, Danderyd Hospital.

Prior to inclusion and randomization, subjects will come at the hospital in order to be subjected to a medical examination, including an electrocardiogram and blood laboratory analyses. Socio-demographic data and medical history will be assessed at this occasion, as well as body variables (weight, height, body composition) and physical activity using the Swedish version of the IPAQ (International Physical Activity Questionnaire). History of major depression will be assessed using the Mini-International Neuropsychiatric Interview (M.I.N.I.) for major depression. Psychological variables that could affect the behavioral (or immune) response to LPS, and which are not believed to change between the screening day and the trial days, will be also assessed at that time, using several web-based self-assessment questionnaires. These measures will include the subjects' perception of the body and health risk (e.g., interoceptive awareness, perceived vulnerability to disease, health anxiety and disgust reactivity, somatosensory amplification, fear of anxiety-related sensations) and psychological well-being (e.g., perceived stress, optimism, social support, cognitive well-being). The overall time for the medical examination will be of 30-45 minutes. The time to complete questionnaires is estimated to approximately 45 minutes but can be done from home. The participants will also receive a kit with a T-shirt (with sewn-in cotton pads) and a scent-free soap. Participants will be asked to wear the T-shirt in the morning (after washing armpits) on each trial day, and take it off after their arrival. This will allow collecting pre-treatment (baseline) samples of body odor.

Participants will then be subjected to the two trials performed in a randomized order, with at least six weeks of wash-out: endotoxin versus placebo.

The participants will be asked to restrain from strenuous exercise and alcohol taking 48 hours before the trial day, to avoid strong spices 24 hours before the trial day, and to take a light breakfast the morning of the trial day. Participants will arrive on the morning (at 7.30AM). They will turn in their morning T-shirt (see above) and change to a new T-shirt (with sewn-in cotton pads in the armpit) to wear during all day. The T-shirts will be used for behavioral assessment and analysis of body odor compound. Shortly after their arrival, two intravenous catheters will be placed: one for blood sampling at one arm and one at one hand for the injection of endotoxin or sodium chloride that will be removed after the injection. An anesthetic cream will be provided to spread on their arm in order to minimize the pain of venipuncture. Subjects will then rest for at least 30 minutes.

Injection of endotoxin or sodium chloride will be performed when the rest is completed (around 8.30AM). Blood samples (10 mL in EDTA (Ethylenediaminetetraacetic acid) tubes and 10 mL in sodium citrate tubes) will be taken just before the endotoxin or sodium chloride injection and 1, 1.5, 2, 3, 4, 5, 6 and 7.5 hours after the injection. In addition, 2.5 mL in PAXGene™ tubes will be taken before and 2, 4 and 7.5 hours after the injection. Two additional samples in EDTA tubes (8 mL of blood) will be taken before the injection and 3 and 7.5 hours after the injection. The total quantity of blood taken will be of about 200 mL, corresponding to a third of the amount given at a blood donation. Blood samples will be used to measure concentrations of pro- and anti-inflammatory cytokines and other inflammatory markers (e.g., C-Reactive protein - CRP) using Enzyme-Linked Immunosorbent Assay (ELISA), immune cell subpopulations and concentrations of microparticles using flow cytometry, genetic markers using Cap analysis gene expression (CAGE) analyses and white blood cell count and differential.

Urine samples will be taken before the endotoxin or sodium chloride injection (i.e., before the catheters are placed) and as late as possible after the injection (classically around four hours after the injection).

Participants will be monitored with continuous electrocardiogram. Oxygen saturation (SO2), blood pressure and body temperature will be monitored every 30 minutes. Nitrogen dioxide (NO2) will be monitored continuously, methemoglobin checked at the same time than each blood sample.

Self-assessment questionnaires assessing behavioral and psychological variables will be completed by participants just before the endotoxin or sodium chloride injection (during the rest period), three hours and 7.5 hours after the injection. A short questionnaire assessing sickness behavior (SicknessQ) will be repeatedly completed by participants from just before to 7.5 hours after the endotoxin or sodium chloride injection. Subjects will be filmed when in bed and will wear a sociometric badge, in order to analyze participants' behavioral response to a standardized situation of social interaction.

Photographs will be taken before (i.e., before the catheters are placed), two hours after and 7.5 hours after the injection, for the further rating of the faces (e.g., health, attractiveness, tiredness). In parallel, skin color will be measured at the same time than blood samples (except T1.5) in order to assess a potential mediating effect of faces' health ratings. Analysis of subjects' gait and motion will be performed two and half hours after the injection. Short computerized cognitive tests will be performed after these tests, just before three hours after the injection. Subjects will perform a motivation task after completing the questionnaires three hours after the injection. In addition, two tests assessing behavior in response to positive/negative and healthy/sickness stimuli (an approach-avoidance behavior test and a regulation of emotion test) will be executed three hours and half after the injection.

Participants will be allowed to take a light meal (snack and juice drink) around lunch time (12.30) and will hand in their T-shirt just before five and half hours after the injection.

The last blood samples will be taken 7.5 hours after the injection and participants will be discharged.

Monitoring of the experiment will be done by a medical doctor, supervised by a specialist in anesthesia and intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diagnosed physiological or psychiatric disease
* Needle anxiety or blood phobia
* Regular medication (excluding contraceptive pill)
* Infection in the last two weeks
* Pregnancy or breastfeeding
* Smoking
* Excessive alcohol use
* Body mass index in the range of obesity (>30 kg/m2) or underweight (<18.5 kg/m2)
* Invisible veins in the antecubital area of the arms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sickness behavior as measured using the sicknessQ | Before the administration and 1.5, 3, 5 and 7 hours after the administration
  Change in sickness behavior evaluated using the self-assessment questionnaire sicknessQ
Change from baseline in anxiety state as measured using the STAI-State | Before the administration and 3 and 7 hours after the administration
  Change in symptoms of anxiety evaluated using the self-assessment questionnaire State part of the State-Trait Anxiety Inventory (STAI)
Change from baseline in psychological state as measured using the SCAS | Before the administration and 3 and 7 hours after the administration
  Change in mood alterations evaluated using the self-assessment questionnaire Swedish Core Affect Scales (SCAS)
Change from baseline in pain as measured using the short McGill questionnaire | Before the administration and 3 and 7 hours after the administration
  Change in symptoms of pain evaluated using the self-assessment questionnaire Mc Gill questionnaire - short version
Change from baseline in sleepiness as measured using the KSS | Before the administration and 3 and 7 hours after the administration
  Change in sleepiness evaluated using the Karolinska Sleepiness Scale (KSS)
Change from baseline in systemic IL-6 concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the pro-inflammatory cytokine interleukin-6 (IL-6)
Change from baseline in systemic TNF-a concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the pro-inflammatory cytokine tumor necrosis factor-alpha (TNF-a)
Change from baseline in systemic IL-8 concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the pro-inflammatory cytokine interleukin-8 (IL-8)
Change from baseline in systemic HMGB1 concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the pro-inflammatory cytokine high-mobility group box 1 (HMGB1)
Change from baseline in systemic IL-1B concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the pro-inflammatory cytokine interleukin-1 beta (IL-1B)
Change from baseline in systemic IL-10 concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the anti-inflammatory cytokine interleukin-10 (IL-10)
Change from baseline in systemic IL-1ra concentrations | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Change in plasma concentration of the anti-inflammatory cytokine interleukin-1 receptor antagonist (IL-1ra)
Change from baseline in heart rate | Before the administration and every half hour up to 7.5 hours after the administration
  Change in heart rate assessed using a cardiac monitoring
Change from baseline in systolic blood pressure | Before the administration and every half hour up to 7.5 hours after the administration
  Change in systolic blood pressure assessed using a cardiac monitoring
Change from baseline in diastolic blood pressure | Before the administration and every half hour up to 7.5 hours after the administration
  Change in diastolic blood pressure assessed using a cardiac monitoring
Change from baseline in body temperature | Before the administration and every half hour up to 7.5 hours after the administration
  Change in body temperature measured using an ear thermometer
Change from baseline in headache scores as measured using a numerical scale | Before the administration and every half hour up to 7.5 hours after the administration
  Change in headache scores measured using a numerical scale ranging from 0 (no headache) to 10 (most unbearable headache)
Change from baseline in nausea scores as measured using a numerical scale | Before the administration and every half hour up to 7.5 hours after the administration
  Change in nausea scores measured using a numerical scale ranging from 0 (no nausea) to 10 (most unbearable nausea)
Change from baseline in back pain scores as measured using a numerical scale | Before the administration and every half hour up to 7.5 hours after the administration
  Change in back pain scores measured using a numerical scale ranging from 0 (no back pain) to 10 (most unbearable back pain)

SECONDARY OUTCOMES:
Change in cell expression of blood microparticles | Before the administration and 1, 1.5, 2, 3, 4, 5, 7 hours after the administration
  Changes in concentrations of total microparticles (defined as particles less than 1μm in size and staining for lactadherin) and platelet-, monocytes- and endothelial-derived microparticles (co-staining of lactadherin and, respectively, cluster of differentiation (CD)42A, CD14 and CD62E).
Modification in genetic markers | Before the administration and 1, 2, 4, 7 hours after the administration
  Modification in genetic markers measured using CAGE analysis from PAXGene blood samples
Change in expression of immune cell markers | Before the administration and 1, 2, 3, 4, 7 hours after the administration
  Change in expression of immune cell subpopulations markers using flow cytometry from frozen whole blood in 10% Dimethylsulfoxid (DMSO)
Change in odor compounds | Before and after the administration
  Change in abundance of volatile odor compounds analyzed using gas chromatography mass spectrometry (GC-MS) from tee-shirt samples and urine samples
Changes in social interaction | During all day
  Modification in social interactions using movies of the study day and sociometric badges
Gait | 2 hours after the administration
  Gait analysis using the Kinect camera
Approach-avoidance behavior | 5 hours after the administration
  Whole-body approach-avoidance behavior to positive/negative stimuli
Face expression of sickness | Before the administration and 2 and 7.5 hours after
  Face expression of sickness measured using photos of the subject with a neutral face expression
Change in skin color | Before the administration and 1,2,3,4,5,7 hours after
  Change in skin color measurement using a spectrophotometer
Motivation as measured using the Effort Expenditure for Rewards Task (EEfRT) | 4 hours after the administration
  Choices of hard task (vs easy task) in the EEfRT

REFERENCES:
- [Derived] Lasselin J, Petrovic P, Olsson MJ, Paues Goranson S, Lekander M, Jensen KB, Axelsson J. Sickness behavior is not all about the immune response: Possible roles of expectations and prediction errors in the worry of being sick. Brain Behav Immun. 2018 Nov;74:213-221. doi: 10.1016/j.bbi.2018.09.008. Epub 2018 Sep 11. PMID 30217536
- [Derived] Axelsson J, Sundelin T, Olsson MJ, Sorjonen K, Axelsson C, Lasselin J, Lekander M. Identification of acutely sick people and facial cues of sickness. Proc Biol Sci. 2018 Jan 10;285(1870):20172430. doi: 10.1098/rspb.2017.2430. PMID 29298938